CLINICAL TRIAL: NCT07215390
Title: A Phase 2, Randomized, Placebo Controlled, Multicenter, Masked Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacodynamics of Multidose APL 3007 in Combination With Syfovre/Pegcetacoplan (APL-2) in Patients Diagnosed With Geographic Atrophy Secondary to Age Related Macular Degeneration
Brief Title: A Phase 2, Randomized, Placebo Controlled, Multicenter, Masked Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacodynamics of Multidose APL 3007 in Combination With Syfovre/Pegcetacoplan (APL-2) in Patients Diagnosed With Geographic Atrophy Secondary to Age Related Macular Degeneratio
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APL3007-GA-201
Record Dates: First submitted 2025-06-30; First posted 2025-10-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-10

CONDITIONS: Geographic Atrophy Secondary to Age-related Macular Degeneration
MeSH Terms: interventions — pegcetacoplan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (APL-3007 Dose/Frequency 1 ) (Experimental): APL-3007 SC + pegcetacoplan (APL-2)
  Interventions: Drug: APL-3007, pegcetacoplan (APL-2)
- Group 2 (APL-3007 Dose/Frequency 2) (Experimental): APL-3007 + pegcetacoplan (APL-2)
  Interventions: Drug: APL-3007, pegcetacoplan (APL-2)
- Group 3 (placebo) (Placebo Comparator): Placebo SC + pegcetacoplan (APL-2)
  Interventions: Other: Placebo, Syfovre

INTERVENTIONS:
Drug: APL-3007, pegcetacoplan (APL-2) — Complement C3 inhibitor
  Arms: Group 1 (APL-3007 Dose/Frequency 1 )
Drug: APL-3007, pegcetacoplan (APL-2) — Complement C3 Inhibitor
  Arms: Group 2 (APL-3007 Dose/Frequency 2)
Other: Placebo, Syfovre — Complement C3 Inhibitor
  Arms: Group 3 (placebo)

SUMMARY:
A Phase 2, Randomized, Placebo-controlled, Multicenter, Masked Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacodynamics of Multidose APL-3007 in Combination with Syfovre/Pegcetacoplan (APL-2) in Patients Diagnosed with Geographic Atrophy Secondary to Age-Related Macular Degeneration

ELIGIBILITY:
Inclusion Criteria:

* The study eye must meet all inclusion criteria. If both eyes meet the inclusion criteria, the eye with better normal luminance visual acuity at the screening visit will be designated as the study eye. If both eyes have the same visual acuity, the right eye will be used as the study eye.
* Aged ≥60 years
* Clinical diagnosis of GA of the macula secondary to AMD in one or both eyes, as determined by the investigator and confirmed by the reading center
* NL-BCVA of 50 letters or better using early treatment diabetic retinopathy study (ETDRS) charts (approximately 20/100 Snellen equivalent)
* Adequate clarity of ocular media, adequate pupillary dilation, and fixation to permit the collection of good quality images in the study eye as determined by the investigator
* Prior treatment for GA in the study eye using Syfovre at 6-8 weeks interval for at least 6 months but no more than 24 months. Participants will be included if the participant has had at least 2 Syfovre injections in the last 6 months before screening.
* The GA lesion in at least 1 eye (designated as the study eye) must meet the following criteria as determined by the central reading center's OCT based RPE assessment of imaging at screening:

  * Total GA area must be ≥2.5 and ≤17.5 mm2 (1-7 disk areas [DA])
  * If GA is multifocal, at least 1 focal lesion must be ≥1.25 mm2 (0.5 DA), with the overall aggregate area of GA as specified above in 7a
  * The entire GA lesion must be completely visualized in the field of view of the OCT, with the GA RPE lesion border >500 µm from the edge of the imaging window or any areas of peripapillary atrophy.
  * Nonsubfoveal lesion with border of GA lesion not encroaching center of the fovea. Distance of GA RPE lesion from center of the fovea >0 based on OCT imaging.
  * Presence of any pattern of hyperautofluorescence based on FAF imaging in the junctional zone of GA. Absence of hyperautofluorescence (ie, pattern = none) is exclusionary.
* Documented evidence of vaccination within 5 years prior to screening, or willing to initiate vaccinations at least 14 days prior to dosing against:

  * Streptococcus pneumoniae (with a pneumococcal conjugate vaccine 15 [PCV15] or 20 [PCV20] or with pneumococcal polysaccharide vaccine 23 [PPSV23]),
  * Haemophilus influenzae (type B) (with Hib vaccine),
  * Neisseria meningitidis types A, C, W, and Y (with a quadrivalent meningococcal conjugate vaccine [eg, Menactra or MenQuadfi]), and
  * Neisseria meningitidis type B (with a meningococcal serogroup B vaccine [eg, Bexsero])

Female participants must be:

* Women of non-childbearing potential (WONCBP), or
* Women of childbearing potential (WOCBP) with a negative serum pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study and refrain from breastfeeding for the duration of the study (see Section 10.9.5.1)

Male participants must be surgically sterile or must agree to use highly effective contraception from screening through the duration of the study

Willing and able to provide informed consent and adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Uncontrolled, clinically relevant history of any gastrointestinal, renal, hepatic, bronchopulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological or allergic disease, metabolic disorder, or cancer
2. History or presence of hepatic cirrhosis or other liver disease that may increase the risk of drug-induced liver injury
3. History or presence of systemic autoimmune disorders, with the exception of well controlled Hashimoto's thyroiditis
4. History of allergy, hypersensitivity, or serious adverse reaction to siRNA therapy or related compounds, or allergy to any of the components of the study drug
5. Clinically meaningful abnormalities on diagnostic and laboratory testing must be adjudicated by the sponsor's medical monitor and include:

   1. Cardiac

      Sustained resting heart rate outside of range of 40 to 100 beats/minute, or a heart rhythm that is not sinus rhythm, confirmed on repeat testing within a maximum of 30 minutes, at screening

      History or evidence of hereditary short QT syndrome

      Fridericia's corrected QT interval (QTcF) >480 milliseconds, or the PR interval outside the range of 120 to 220 milliseconds, confirmed on repeat testing within a maximum of 30 minutes at screening

      Any clinically relevant features of acute coronary syndrome (unstable angina, myocardial infarction)

      Any other ECG parameters outside of age-adjusted normative range
   2. Hepatic

      AST or ALT >1.3 × ULN

      Total bilirubin >1.1 × ULN

      Any 2 LFTs >1.1 × ULN

      Any other LFT parameters outside of age-adjusted normative range
   3. Renal

   Estimated glomerular filtration rate of less than <45 mL/min/m2 as calculated by the Chronic Kidney Disease-Epidemiology Collaboration (CKD- EPI) creatinine equation for adults

   Any other renal function parameters outside of age-adjusted normative range
6. History or presence of malignancy (except history of basal or squamous cell carcinoma of the skin) that has not been successfully treated ≥1 year prior to enrollment
7. History or presence of recurrent or unexplained infections, HIV infection, hepatitis B, hepatitis C, or meningococcal infection
8. Participants with fever (defined as temperature >100.4 °F/38 °C) or any acute infection (including COVID-19 infection or infection requiring antibiotic treatment) within 30 days of screening until dosing
9. Evidence of ongoing drug or alcohol abuse or dependence, in the opinion of the investigator
10. Intention to donate sperm during this study or within 90 days after the last dose of study drug
11. Prior administration of APL-3007
12. Participation in an investigational product or medical device study within 5 half-lives of the investigational product before the screening visit
13. Has poor peripheral venous access or any abnormal skin conditions or potentially obscuring tattoos, pigmentation, or lesions in the area intended for SC injection that would interfere with SC injections or assessments of injection local tolerability
14. Any condition which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the investigator or medical monitor(s), unacceptably increase the participant's risk by participating in the study
15. Has received a live vaccination (excluding seasonal flu vaccination) within 30 days prior to the first dose administration
16. Women who are pregnant or breastfeeding
17. Medical or psychiatric conditions that, in the opinion of the investigator, make consistent follow-up over the treatment period unlikely, or would make the participant an unsafe study candidate

    Ocular specific exclusion criteria apply to the study eye only, unless otherwise specified.
18. GA secondary to a condition other than AMD such as Stargardt disease, cone rod dystrophy or toxic maculopathies like plaquenil maculopathy in either eye
19. Any history of CNV (active or nonexudative/quiescent) in the study eye associated with AMD or any other cause, including any evidence of RPE rips, double layer sign, or evidence of neovascularization anywhere based on SD-OCT imaging and fluorescein angiography as assessed by the reading center
20. Presence of an active ocular disease that, in the opinion of the investigator, compromises or confounds visual function, including but not limited to, uveitis, other macular diseases (eg, clinically significant epiretinal membrane, full thickness macular hole or uncontrolled glaucoma/ocular hypertension); benign conditions in the opinion of the investigator such as peripheral retina dystrophy are not exclusionary.
21. History of IVT injection in the study eye within 3 months prior to the screening visit, with the exception of IVT Syfovre
22. History of any previous investigational product for GA treatment in either eye within 3 months (or 5 half-lives of the investigational drug, whichever is longer) prior to the screening visit
23. History of laser therapy in the macular region
24. Any ocular condition other than GA secondary to AMD that may require surgery or medical intervention during the study period or, in the opinion of the investigator, could compromise visual function during the study period

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline (CFB) in the area of artificial intelligence (AI)-based SD-OCT assessment of RPE lesion in the study eye | At month 12

SECONDARY OUTCOMES:
CFB in the area of AI-based OCT assessment of photoreceptor degeneration in the study eye | At month 12
Safety & tolerability based on adverse event (AE) reporting | At month 12
Safety as assessed by Best Corrected Visual Acuity (BCVA) | At Month 12
  Continuous monitoring of a subject' BCVA as assessed by EDTRS chart
Change from baseline in Serum C3 level | At Month 12
  Continuous monitoring of a subject's Serum C3 level
CFB in RPE lesion area as assessed by FAF in the study eye | At month 12
CFB in the junctional zone, central 2o and 6o MP number of scotomatous points in the study eye | At month 12
CFB in the junctional zone, central 2o and 6o MP mean sensitivities in the study eye | At month 12
CFB in normal luminance qCSF in the study eye as assessed with the Adaptive Sensory Technology Manifold Platform | At month 12
CFB in low luminance qCSF in the study eye as assessed with the Adaptive Sensory Technology Manifold platform | At month 12

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Associated Retina Consultants - Phoenix, Phoenix, Arizona
  - California Retina Consultants (CRC) - Bakersfield Office, Bakersfield, California
  - The Retina Partners - Encino, Encino, California
  - Retina Consultants of Orange County - Fullerton Office, Fullerton, California
  - Retina Consultants San Diego, Poway, California
  - Bay Area Retina Associates - Walnut Creek, Walnut Creek, California
  - Advanced Vision Research Institute, Longmont, Colorado
  - Retina Specialty Institute - Pensacola, Pensacola, Florida
  - Retina Vitreous Associates of Florida (RVA) - Saint Petersburg, St. Petersburg, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Cumberland Valley Retina Consultants (CVRC), Hagerstown, Maryland
  - Mississippi Retina Associates, Madison, Mississippi
  - Long Island Vitreoretinal Consultants - Westbury, Long Island City, New York
  - Verum Research, LLC, Eugene, Oregon
  - EyeHealth Northwest, Portland, Oregon
  - Charleston Neuroscience Institute LLC - Ladson, Ladson, South Carolina
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas - Katy, Katy, Texas
  - Retina Consultants of Texas - San Antonio Medical Center, San Antonio, Texas
  - Retina Consultants of Texas - The Woodlands, The Woodlands, Texas
  - Tyler Retina Consultants, Tyler, Texas
  - University of Wisconsin Health - University Station Clinic, Madison, Wisconsin